CLINICAL TRIAL: NCT03764358
Title: Comparison of Tunneled Cuffed Dialysis Catheters Versus Arteriovenous Fistulae in Elderly or Multimorbid Patients
Brief Title: AUSTrian Randomized Interventional Study on Dialysis Accesses
Acronym: AUSTRIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Guerkan SENGOELGE, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AUSTRIA
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: End Stage Renal Disease; Catheter Infection; Shunt Malfunction
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Arteriovenous Shunt, Surgical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arteriovenous fistula (Active Comparator)
  Interventions: Device: Arteriovenous Fistula
- Tunneled Cuffed Catheter (Experimental)
  Interventions: Device: Tunneled Cuffed Catheter

INTERVENTIONS:
Device: Arteriovenous Fistula — Surgical implantation of an arteriovenous fistula for hemodialysis
  Arms: Arteriovenous fistula
Device: Tunneled Cuffed Catheter — Placement of a tunneled cuffed catheter in surgical theatre
  Arms: Tunneled Cuffed Catheter

SUMMARY:
Patients with diagnosed end stage renal disease and indication for chronic dialysis rely on a well-functioning access for dialysis. The KDOQI Guidelines For Vascular Access follows a "fistula first" approach for every patient, whenever possible. Thus, every patient, regardless of age, clinical state and co-morbidities an arteriovenous fistula should be preferred over a tunneled cuffed catheter (TCC). These recommendations are based on retrospective and register studies. There have been no prospective studies in this subject so far. In addition, most of the collected data refers to patients of all ages, regardless of their comorbidities and general clinical state. In this study, we address differences between two dialysis vascular access types in elderly or frail patients. We will compare TCCs with arteriovenous fistulas in the selected population consisting of elderly patients over 60 years of age or those with a Charlson Comorbidity Index >6 independent of age. In our hypothesis TCCs will be superior to arteriovenous fistulas in this population regarding the examined end-points.

ELIGIBILITY:
Inclusion Criteria:

* Age of 60 and higher
* CCI Score >6 when under 60 years
* Patients with CKD G5 A1-3 with indication for hemodialysis
* Stable clinical condition
* Eligibility for both arteriovenous fistula on the upper extremitiesandTCC
* Availability for follow-up.
* Written informed consent.

Exclusion Criteria:

* Uncontrolled infection at screening and/or CRP >5 mg/dl (normal <0.5 mg/dl) at screening.
* Poor general condition of health or malignancy not in remission at screening
* Major surgery within 12 weeks before screening.
* Pre-existent vascular access.
* Patient not eligible for any one of the vascular access options.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-03-06 (Estimated); Primary Completion 2022-04-04 (Estimated); Study Completion 2022-10-04 (Estimated)

PRIMARY OUTCOMES:
Composite primary end-point of any access related complication | From placement of vascular access through study completion, an average of 3 years.
  Loss of access, catheter related bloodstream infection/shunt infection and/or thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Guerkan Sengoelge, MD, Principal Investigator — Medical University of Vienna, Department of Medicine III, Devision of Nephrology and Dialysis
Locations (1):
- Department of Medicine III, Devision of Nephrology and Dialysis, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided